CLINICAL TRIAL: NCT01859117
Title: A Phase 1 Multicenter, Open-Label, Dose-Escalation Study to Evaluate the Safety and Efficacy of Intramuscular Injection of Human Placenta-Derived Cells (PDA-002) in Subjects With Peripheral Arterial Disease and Diabetic Foot Ulcer
Brief Title: Study of Human Placenta-derived Cells (PDA002) to Evaluate the Safety and Effectiveness in Subjects With PAD and DFU
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celularity Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCT-PDA-002-DFU-001
Record Dates: First submitted 2013-05-17; First posted 2013-05-21 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2017-02

CONDITIONS: Peripheral Arterial Disease; Diabetic Foot
Keywords: Peripheral arterial disease; diabetic foot
MeSH Terms: conditions — Peripheral Arterial Disease; Diabetic Foot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 3 x 10^6 cells (Experimental): 3 x 10^6 Human Placenta Derived cells (PDA-002) administered intramuscularly on Study Days 1 and 8
  Interventions: Biological: 3 x 10^6 cells
- 10 x 10^6 cells (Experimental): 10 x 10^6 Human Placenta Derived cells (PDA-002) administered intramuscularly on Study Days 1 and 8
  Interventions: Biological: 10 x 10^6 cells
- 30 x 10^6 cells (Experimental): 30 x 10^6 Human Placenta Derived cells (PDA-002) administered intramuscularly on Study Days 1 and 8
  Interventions: Biological: 30 x 10^6 cells
- 100 x 10^6 cells (Experimental): 100 x 10^6 Human Placenta Derived cells (PDA-002) administered intramuscularly on Study Days 1 and 8
  Interventions: Biological: 100 x 10^6 cells

INTERVENTIONS:
Biological: 3 x 10^6 cells — 3 x 10^6 cells administered on Study Days 1 and 8
  Other Names: PDA-002
  Arms: 3 x 10^6 cells
Biological: 10 x 10^6 cells — 10 x 10^6 cells administered on Study Days 1 and 8
  Other Names: PDA-002
  Arms: 10 x 10^6 cells
Biological: 30 x 10^6 cells — 30 x 10^6 Human Placenta Derived cells (PDA-002) administered intramuscularly on Study Days 1 and 8
  Other Names: PDA-002
  Arms: 30 x 10^6 cells
Biological: 100 x 10^6 cells — 100 x 10^6 cells administered on Study Days 1 and 8
  Other Names: PDA-002
  Arms: 100 x 10^6 cells

SUMMARY:
This clinical study is being conducted to assess the safety and determine the maximum tolerated dose (MTD) of PDA-002 [human placenta-derived cells] administered into the lower leg muscles of subjects with peripheral arterial disease and diabetic foot ulcers. It will look to see if PDA-002 helps reduce some of the symptoms of PAD and/or improves ulcer healing. This study will also help to find the best dose of PDA-002 to use in future studies.

DETAILED DESCRIPTION:
The goal of this study is to determine a safe dose of PDA-002 [human placenta-derived cells] for further study. This is a dose-escalation study where each of four dose levels will enroll three to six subjects. Doses will be range from 3 million up to 100 million cells. If one dose is considered safe after all treated subjects have been evaluated and reviewed, then the next group of subjects will be enrolled to receive the next higher dose. This will continue until either the highest dose is reached, until at least 2 subjects at a dose level have ≥ Grade 2 allergic reaction that is suspected to be related to PDA-002 or 2 or more subjects at a dose level experience an unexpected, treatment-related serious adverse event or dose limiting toxicity within 14 days following the initial dose of PDA-002. This is an open-label study where all subjects will be taking the study drug and all study personnel will know the dose each subject receives.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must satisfy the following criteria to be enrolled in the study:

  1. Males and females, 18 to 80 years of age at the time of signing the informed consent document.
  2. Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures are conducted.
  3. Able to adhere to the study visit schedule and other protocol requirements.
  4. Diabetes mellitus type 2
  5. Ischemic or neuro-ischemic diabetic foot ulcer with severity of Grade 1 (full thickness only) or Grade 2 on the Wagner Grading Scale (Appendix A) of greater than one month duration which has not adequately responded to conventional ulcer therapy.
  6. Peripheral arterial disease with ankle-brachial index > 0.6 and ≤ 0.9 or toe-brachial index > 0.35 and ≤ 0.7.
  7. No planned revascularization or amputation over the next 3 months after Screening visit, in the opinion of the Investigator.
  8. Not a candidate for peripheral artery percutaneous or surgical revascularization.
  9. Screening should not begin until at least 2 weeks after a failed reperfusion intervention and at least 2 months after a successful mechanical intervention.
  10. Subject can have stable angina, (Canadian Cardiovascular Society (CCS) Class I-II angina (Appendix H).
  11. Subjects should be receiving appropriate medical therapy for hypertension and diabetes.
  12. Subject must be a non-tobacco user defined as someone who has not used tobacco/nicotine patch for ≥ 3 months and must agree to remain tobacco/nicotine free for the duration of the study.
  13. A female of childbearing potential [FCBP] must have a negative serum pregnancy test at Screening and a negative urine pregnancy test prior to treatment with study therapy. In addition, sexually active FCBP must agree to use 2 of the following adequate forms of contraception methods simultaneously such as: oral, injectable, or implantable hormonal contraception; tubal ligation; intrauterine device [IUD]; barrier contraceptive with spermicide or vasectomized partner for the duration of the study and the follow-up period.
  14. Males (including those who have had a vasectomy) must agree to use barrier contraception (latex condoms) when engaging in reproductive sexual activity with FCBP for the duration of the study and the follow-up period.

      Exclusion Criteria:
* The presence of any of the following will exclude a subject from enrollment:

  1. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
  2. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he or she were to participate in the study.
  3. Any condition that confounds the ability to interpret data from the study.
  4. Subjects whom, in the judgment of the Investigator, are at elevated risk for the development of a malignancy. This judgment may be based on family history, history of industrial exposures, smoking history or other cancer risk factors.
  5. Known to be positive for human immunodeficiency virus.
  6. Pregnant or lactating females.
  7. Subjects with a body mass index > 35 at Screening.
  8. Aspartate transaminase (AST) or Alanine transaminase (ALT) > 2.5 x the upper limit of normal (ULN) at Screening.
  9. Estimated Glomerular Filtration Rate (eGFR) < 45 mL/min/1.73 m2 at Screening calculated using the Modification of Diet in Renal Disease Study equation (Levey, 2006) or history of eGFR decline > 15 mL/min/1.73 m2 in the past year.
  10. Alkaline phosphatase > 2.5 x the ULN at Screening.
  11. Bilirubin level > 2 mg/dL (unless subject has known Gilbert's disease) at Screening.
  12. Untreated chronic infection or treatment of any infection with systemic antibiotics, including the ulcer site, within 4 weeks prior to dosing with investigational product [IP].
  13. Known osteomyelitis.
  14. History of Methicillin-resistant Staphylococcus aureus (MRSA).
  15. Ulcer that has decreased or increased in size by ≥ 50% during the screening period.
  16. Uncontrolled hypertension (defined as diastolic blood pressure > 100 mmHg or systolic blood pressure > 180 mmHg during Screening at 2 independent measurements taken while subject is sitting and resting for at least 5 minutes).
  17. Poorly controlled diabetes mellitus (hemoglobin A1c > 9%).
  18. Untreated proliferative retinopathy.
  19. History of malignant ventricular arrhythmia, CCS Class III-IV angina pectoris, myocardial infarction/PCI (percutaneous coronary intervention)/CABG (coronary artery bypass graft) in the preceding 6 months, pending coronary revascularization in the following 2 months, transient ischemic attack/cerebrovascular accident in the preceding 6 months, and/or New York Heart Association [NYHA] Stage III or IV congestive heart failure, (Appendix C).
  20. Abnormal ECG: new bundle branch block (BBB) ≥ 120 msec in the preceding 3 months; QTcB and/or QTcF > 480 msec or QTcB and/or QTcF ≥ 500 msec with old BBB. Patients with a potential risk for Torsades des Pointes should not be enrolled.
  21. Uncontrolled hypercoagulation.
  22. Life expectancy less than 2 years due to concomitant illnesses.
  23. In the opinion of the Investigator, the subject is unsuitable for cellular therapy.
  24. History of malignancy within 5 years except basal cell or squamous cell carcinoma of the skin or remote history of cancer now considered cured or positive Pap smear with subsequent negative follow-up.
  25. History of hypersensitivity to any of the components of the product formulation (including bovine or porcine products, dextran 40, and dimethyl sulfoxide [DMSO]).
  26. Disorders or allergies precluding the use of radiographic contrast or renal insufficiency severe enough to contraindicate the use of radiographic contrast.
  27. Subject has received an investigational agent -an agent or device not approved by the US Food and Drug Administration (FDA) for marketed use in any indication- within 90 days (or 5 half-lives, whichever is longer) prior to treatment with study therapy or planned participation in another therapeutic study prior to the completion of this study.
  28. Subject has received previous gene or cell therapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 14 days of initial dosing
  To determine the maximum tolerated dose (MTD) of PDA-002 administered intramuscularly (IM) in subjects with peripheral arterial disease (PAD) and DFU [diabetic foot ulcer].
Adverse Events | From signing informed consent until month 24
  Number of participants with adverse events

SECONDARY OUTCOMES:
Ankle-brachial index (ABI) | Approximately 2 years
  at the ankle by the systolic blood pressures (Doppler technique) in the arm.
Toe-brachial index (TBI) | Approximately 2 years
  To assess changes in the TBI which is calculated by dividing the systolic blood pressure at the toe by the systolic blood pressures (Doppler technique) in the arm.

CONTACTS AND LOCATIONS:
Overall Officials: Monica E Luchi, MD, Study Director — Celularity Incorporated
Locations (11):
- United States (11):
  - Carl T. Hayden Veterans Affairs Medical Center, Phoenix, Arizona
  - UCLA, Los Angeles, California
  - Stanford University School of Medicine, Stanford, California
  - Dr. Wiliam M. Scholl College of Podiatric Medicine, North Chicago, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - University of North Carolina School of Medicine, Chapel Hill, North Carolina
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Complete Family Foot Care - McAllen Office, McAllen, Texas
  - Endeavor Clinical Trials PA, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - University of Wisconsin, Madison, Wisconsin

REFERENCES:
- [Derived] Francki A, Labazzo K, He S, Baum EZ, Abbot SE, Herzberg U, Hofgartner W, Hariri R; Celgene Cellular Therapeutics Research Group. Angiogenic properties of human placenta-derived adherent cells and efficacy in hindlimb ischemia. J Vasc Surg. 2016 Sep;64(3):746-756.e1. doi: 10.1016/j.jvs.2015.04.387. Epub 2015 Jun 6. PMID 26054585